CLINICAL TRIAL: NCT02511002
Title: Long-Term Observation of Hemagglutinin and Neuraminidase Inhibition Antibody Titers After Influenza Challenge
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150154; 15-I-0154
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-10

CONDITIONS: Post Influenza
Keywords: Natural History; Longitudinal Observation; Influenza Like Infection (ILI); Immunity; Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Post influenza infection

SUMMARY:
Background:

- Influenza is a common viral infection, but it can be deadly for some people. Researchers want to learn more about how the body fights this virus. They want to study this in people who have recently been infected with influenza. They hope this can help them create more effective influenza vaccines.

Objective:

- To learn about long-term changes in the body s immune system after influenza infection.

Eligibility:

- People who have completed a previous LID Clinical Studies Unit influenza challenge study or current or prior participation in an LID natural history study and are willing to have samples stored for future research.

Design:

* Eligible participants will be asked to visit the clinic every 3 months for 2 years.
* During each visit, participants will have blood drawn from an arm vein using a needle and a syringe and a nasal sample.
* Participants will have a medical history and physical exam and vital signs performed. This will include blood pressure, heart rate, breathing rate, temperature, weight, and finger-measured blood oxygen. They will answer questions about any medicines taken and possible recent illnesses.
* If participants have symptoms of influenza, they may have an additional sample taken from the nose.
* Participants will complete a health questionnaire once a month on a secure website. Participants may also give their responses over the telephone....

DETAILED DESCRIPTION:
Circulating anti-influenza antibodies are an important factor in predicting clinical illness and severity in those infected with influenza. Specific antibodies against influenza include proteins targeting hemagglutinin (HA) and neuraminidase (NA). Lifelong immunity does not occur with influenza, either from natural infection or from vaccination. Due to the antigenic variation of Influenza A, individuals may become infected multiple times with the same subtype of influenza and even with the same strain. In the setting of natural infection and vaccination, antibody titer levels can persist initially, but then wane over time.

In our previous challenge studies, measurements of antibody responses have been focused solely on the acute infection period up to 2 months after initial infection. Long-term changes in immunity have not been investigated. The challenge setting gives us the unique ability to follow individuals from a specific, known and well-characterized exposure/illness to measure long-term changes in antibody titers from a pre-exposure baseline. This study could offer unique insight into how anti-influenza antibody titers change over time naturally and in response to other infections and life events. This type of controlled study has never been done and we believe monitoring titers long-term will help us better understand protective correlates of influenza.

In this natural history study, we will follow individuals who have undergone influenza challenge or have been naturally infected with influenza to evaluate changes in anti-influenza antibody titers over a 2-year period. Subjects will be followed for symptoms of influenza-like illness (ILI) and other changes in clinical status through quarterly clinical evaluations with blood draws. Monthly questionnaires will be used to follow subjects in between visits.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Completion of participation in an LID Clinical Studies Unit influenza challenge study or current or prior participation in an LID natural history study.
  2. Willing to have samples stored for future research.

CO-ENROLLMENT GUIDELINES:

Participants may be co-enrolled in other research studies. This will be addressed on a case-by-case basis with the approval of the principal investigator (PI) or associate investigator.

If a participant enrolls in another influenza challenge study, the participant will be removed from this study. The participant can re-enroll in this study after completion of the influenza challenge study and will be followed for two years following completion of the most recent influenza challenge study.

EXCLUSION CRITERIA:

Any condition or event that, in the PI s opinion, may substantially increase the risk associated with study participation or compromise the study s scientific objectives. Conditions that exclude a subject are considered to be unlikely, but an example would include a newly diagnosed medical condition that may alter a participant s immune system and make it unsafe to obtain scheduled blood samples for research purposes.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers after influenza challenge and patients after natural influenza infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07-17 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the timing of peak antibody response to hemagglutinin (HA) and neuraminidase (NA) post influenza challenge or after natural infection To evaluate the long-term variability of hemagglutinin inhibition (HAI) and neuraminidase inhib... | 2 years
  Trend of HAI titer over multiple time points Trend of NAI titer over multiple time points

SECONDARY OUTCOMES:
To correlate changes in clinical status such as influenza-like illness (ILI) or vaccinations with changes in antibody titers and other immune measures | 2 years
  Change in HAI titer before and after change in clinical status Change in NAI titer before and after change in clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Alison Han, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grohskopf LA, Olsen SJ, Sokolow LZ, Bresee JS, Cox NJ, Broder KR, Karron RA, Walter EB; Centers for Disease Control and Prevention. Prevention and control of seasonal influenza with vaccines: recommendations of the Advisory Committee on Immunization Practices (ACIP) -- United States, 2014-15 influenza season. MMWR Morb Mortal Wkly Rep. 2014 Aug 15;63(32):691-7. PMID 25121712
- [Background] Thompson WW, Weintraub E, Dhankhar P, Cheng PY, Brammer L, Meltzer MI, Bresee JS, Shay DK. Estimates of US influenza-associated deaths made using four different methods. Influenza Other Respir Viruses. 2009 Jan;3(1):37-49. doi: 10.1111/j.1750-2659.2009.00073.x. PMID 19453440
- [Background] Cox RJ. Correlates of protection to influenza virus, where do we go from here? Hum Vaccin Immunother. 2013 Feb;9(2):405-8. doi: 10.4161/hv.22908. Epub 2013 Jan 4. PMID 23291930
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-I-0154.html